CLINICAL TRIAL: NCT06205940
Title: Building Individual and Community Resilience Through Nature-based Therapies - Case Study 8
Brief Title: Building Individual and Community Resilience Through Nature-based Therapies - Case Study 8 Nature for All
Acronym: RESONATE-CS8
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 101081420
Record Dates: First submitted 2024-01-03; First posted 2024-01-16 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Mobility Disability
Keywords: nature app; nature connection; forest walks; mobility disability; resilience; eyetracking

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audio guided nature tour (Experimental): Listening to audio instructions by an app while visiting nature.
  Interventions: Behavioral: Audioguided Nature tour
- Non audio guided nature tour (Active Comparator): Visiting nature without audio guided instructions (app).
  Interventions: Behavioral: Non audio guided nature tour

INTERVENTIONS:
Behavioral: Audioguided Nature tour — Listening to audio instructions by an app while visiting nature. The instructions emphasize the connection between self and nature and direct attention to the present moment experience by guiding focus towards sensory experiences and specific natural elements.
  Arms: Audio guided nature tour
Behavioral: Non audio guided nature tour — Visiting nature without listening to audio instructions by an app
  Arms: Non audio guided nature tour

SUMMARY:
The aim of this randomized controlled trial is to test if digital engagement instructions (a nature guide APP) can enhance the nature connection and provide positive health outcomes for individuals with mobility disabilities.

The study has an active control group, that will have the same nature exposure without the guidance of the APP. 124 participants will be randomized to either the intervention group or the control group.

The intervention consists of two parts:

Intervention day 1: The intervention starts for both the 'intervention group' and the 'control group' in the Hoersholm arboretum, which contain Denmark's largest collection of different trees and shrubs. The intervention group will listen to the 'intervention APP' during a tour with three stops along a trail in the arboretum. The active control group will take the same tour but does not have access to the 'intervention APP'.

4 week intervention: During the following 4 weeks the participants will be encouraged to visit nature for 120 minutes in total per week on their own. The intervention group will still be encouraged to use the APP during the nature visits.

DETAILED DESCRIPTION:
See protocol

ELIGIBILITY:
Inclusion Criteria:

* Not being able to walk at all or be able to walk short distances (ICF 2017: d4500, walking short distances; walking for less than a kilometer, such as walking around rooms or hallways, within a building or for short distances outside)
* All types of assistive devices, including e.g. scooters, walkers, and canes. Also service dogs and personal carers are included.
* Adults (+18 years)
* All genders
* All educational levels
* All religious affiliations
* All types of marital status
* All types of households
* All types of employment and income

Exclusion Criteria:

* - Do not understand Danish (APP, questionnaires and interviews in Danish)
* Physically not able to use a smartphone with touch screen, by themselves or with the help of a personal carer
* Participating in mindfulness program during intervention (intervention day 1 and 4-week intervention period)
* Cognitive limitations (difficulties in understanding and using information from APP, understanding and responding to questionnaires and interviews.)
* Known drug or alcohol abuse
* Diagnosed epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
The Nature Connection Index | Baseline 0 (1 week before intervention), After intervention day 1, End of intervention (after 4 months), 1 month follow-up, 3 month-follow up, 6-months follow-up
  Questionnaire Nature Connection Index (NCI) is a 6-item self-report measure of connection to nature. The level of agreement with each of the 6 statements is rated on a scale from 1 (completely agree) to 7 (completely disagree), where a higher score indicates higher level of nature connection.

SECONDARY OUTCOMES:
the State Mindfulness Scale | Baseline 1 (just before intervention), After tour on intervention day 1, End of intervention (after 4 months)
  The State Mindfulness Scale (SMS) is a 21-item self-report measure of state mindfulness. The level of agreement with each of the 21 statements is rated on a scale from 1 (not at all) to 5 (very much), where a higher score indicates higher level of state mindfulness.
The Restorative Outcome Scale | After tour on intervention day 1, End of intervention (after 4 months)
  The Restorative Outcome Scale (ROS) is a 6-item self-report measure of the restorative effect of natural environments. The level of agreement with each of the six statement is rated on a 7 point scale from 0 (completely disagree) to 6 (completely agree), where a higher score indicates higher level of self perceived restorative outcome.
The Subjective Vitality Scale | Baseline 0 (1 week before intervention), After intervention day 1, End of intervention (after 4 months), 1 month follow-up, 3 month-follow up, 6-months follow-up
  The Subjective Vitality Scale (SVS) is a 6-item self-report measure of subjective vitality. The level of agreement with each of the six statement is rated on a 7 point scale from 1(completely disagree) to 7 (completely agree), where a higher score indicates higher level of subjective vitality.
The State-Trait Assessment of Resilience Scale | Baseline 0 (1 week before intervention), After intervention day 1, End of intervention (after 4 months), 1 month follow-up, 3 month-follow up, 6-months follow-up
  The State-Trait Assessment of Resilience Scale (STARS) is a 7-item self-report measure of resilience. The level of agreement with each of the 7 statements is rated on a 4 point scale from 1(disagree) to 4 (completely agree). Item 3,4,5 have reverse scoring. A higher score indicates higher level of subjective vitality.
Heart Rate Variability | During tour on intervention day 1
  HRV analysis will be performed on electrocardiograms, ECG signals
The Health-related Quality of Life Short Form Survey | Baseline 0 (1 week before intervention), End of intervention (after 4 months), 1 month follow-up, 3 month-follow up, 6-months follow-up
  The Health-related Quality of Life Short Form Survey (SF-12) is a 12-item Short Form Survey measuring health related quality of life. Each question is answered on a 6 point scale ranging from not at all (1) to all the time (6). A higher total score indicates higher level of health-related quality of life.

OTHER OUTCOMES:
Eye-tracking | During tour on intervention day 1
  Portable eye-tracking recording
System Usability Scale | After tour on intervention day 1
  The System Usability Scale (SUS) consists of 10 question, scored on a 5 point likert scale ranging from strongly disagree (0) to strongly agree (4), where item 2,4,6,8 and 10 have reverse scoring. A higher score indicate higher level of perceived usability.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika K Stigsdotter, PHD, Principal Investigator — University of Copenhagen - IGN

IPD SHARING:
Plan to Share IPD: Yes
Data is shared exclusively in pseudonymized form with all partners in the RESONATE project. The countries included in RESONATE are: Denmark, Spain, Italy, Belgium, Sweden, Bulgaria, Austria, and the Netherlands. The UK is an associated partner.
Time Frame: 2025 to 2028
Access Criteria: The RESONATE project is currently developing a Joint Control Agreement which is an arrangement on shared responsibility for data processing, which determines in a transparent manner the partner's respective responsibilities for GDPR compliance. Signing this agreement allows results to be shared freely within the consortium. Thus, the RESONATE partners would not need separate Data Sharing or Data Transfer agreements with each partner.
  The General Data Protection Regulation (GDPR) is enforced in all EU countries and also in the UK. All partners in the consortium need to follow the GDPR.